CLINICAL TRIAL: NCT02358668
Title: A Study to Evaluate the Effect of BTI320 (SUGARDOWN®) on Post-Prandial Hyperglycaemia in High Risk Chinese Subjects With Pre-Diabetes
Brief Title: BTI320 (SUGARDOWN®) on Post-Prandial Hyperglycaemia in Subjects With Pre-Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Sugardown Company Limited (Industry)
Responsible Party: Principal Investigator, Andrea On Yan Luk, Assocoiate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG01
Record Dates: First submitted 2015-01-30; First posted 2015-02-09 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Pre-Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — PAZ320

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BTI320 4 grams (Experimental): three times daily, oral for 16 weeks
  Interventions: Drug: BTI320
- BTI320 8 grams (Experimental): three times daily, oral for 16 weeks
  Interventions: Drug: BTI320
- BTI320 matching placebo (Placebo Comparator): 2 tablets three times daily, oral for 16 weeks
  Interventions: Drug: BTI320 matching placebo

INTERVENTIONS:
Drug: BTI320 — BTI320, also known as SUGARDOWN®, is derived from galactomanan which blocks key enzymes that break down carbohydrate in the gut. BTI320 therefore helps to slow down the absorption of carbohydrates to lower post-meal blood sugar.
  Other Names: SUGARDOWN®
  Arms: BTI320 4 grams; BTI320 8 grams
Drug: BTI320 matching placebo — Placebo
  Arms: BTI320 matching placebo

SUMMARY:
This is a single-centre, 16-week, randomized, double-blind, placebo-controlled, 3-treatment arm pilot study to evaluate the efficacy and safety of BTI320 in the treatment of high risk subjects with pre-diabetes.

This is a pilot study aiming to test whether taking a medicine named BTI320 that slows down carbohydrate absorption in the gut, will lower blood sugar. The study aims to recruit 60 individuals in Hong Kong. To take part in the study, subjects must have pre-diabetes, that is, they have blood sugar levels that are above normal but not reaching diabetes range. The medicine BTI320 is currently licensed as a health supplement in Hong Kong and is known alternatively as SUGARDOWN®. The investigators are comparing the effectiveness of BTI320 against a dummy tablet. Both tablets look and taste identical and during the study, subjects will not know which of these tablets they are taking. There is a 4 in 5 chance of receiving active medication and 1 in 5 chance of receiving placebo. Subjects will be followed up closely every 2 to 4 weeks for a period of time up to 22 weeks.

The study visits will take between 30 minutes to 3 hours, depending on additional checks that are required on a particular visit including oral glucose tolerance test and meal tolerance test. At visits involving meal tolerance test, subjects will be required to stay for approximately 3 hours. In addition, at Visit 2, Visit 4 and 3 days before Visit 7, a continuous glucose monitoring system device will be installed.

Throughout the study period, subjects will return to the study center for check-ups including careful enquiry about whether they have developed any side-effects from taking the medication, physical examination, as well as blood tests.

DETAILED DESCRIPTION:
In a recent national survey, 11% of adults in China have diabetes and 50% have pre-diabetes defined by fasting plasma glucose (FPG) 5.6-6.9 mmol/l and/or 2-hour post glucose (PG) 7.8-11.0 mmol/L using 75 gram oral glucose tolerance test (75g OGTT) and/or glycated haemoglobin (HbA1c) 5.7-6.4%. Depending on the presence of other risk factors, the annual conversion rate of pre-diabetes averages 3-10% with pre-diabetes associated with 1.5-2.0 fold increased risk for cardiovascular disease. Once diabetes is established, life expectancy is reduced by 6 years if not diagnosed, treated or controlled, especially in young-to-middle aged subjects who will face long disease duration of diabetes.

In the Hong Kong Diabetes Registry, depending on control of glucose and other risk factors, 3-10% of Chinese subjects with diabetes may die or develop a major event every year including heart disease, stroke, kidney failure and /or all-site cancer.

Besides glycaemic control as defined by HbA1c, post prandial hyperglycaemia and glycaemic variability have also been shown to predict cardiovascular and renal events in both pre-diabetic and diabetic patient. Genetic variants discovered in large-scale epidemiological studies including those from China and Hong Kong have been found to be associated with beta cell dysfunction which can be further exacerbated by glucotoxicity and lipotoxicity, often due to co-existing obesity giving rise to early onset diabetes. Several studies including those from Asian populations indicated that subjects with pre-diabetes exhibit reduced early phase insulin secretion resulting in postprandial hyperglycaemia which can impose metabolic stress on the beta cells leading to eventual beta cell failure.

BTI320, also known as SUGARDOWN®, is derived from galactomanan which acts by blocking the key carbohydrate hydrolyzing enzymes including amylase, maltose, lactose and sucrose in the gastrointestinal tract. It also acts to bind to ingested polysaccharides and slow their absorption with each meal thereby reducing post prandial glucose excursion. The mechanism of action for BTI320 is similar to Acarbose®, an alpha glucosidase inhibitor, which has been shown to improve glycaemic control and has been approved for prevention of diabetes in China.

24-hour continuous glucose monitoring system (CGMS) measures mean blood glucose (MBG), mean area under the curve for blood glucose above 10mmol/l (180mg/dl) (AUC-180), mean postprandial maximum glucose (MPMG), mean amplitude of glucose excursion (MAGE) over 72 hours. These parameters correlate well with plasma fructosamine (FA) alternatively known as glycated albumin, which reflects short-term glycaemic control during the preceding 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects ≥ 18-70 years inclusive
2. Chinese ethnicity
3. High risk subject with pre-diabetes as defined by meeting at least 2 of the following criteria from (a), (b) and (c):

   1. FPG ≥ 5.6-6.9 mmol/l and/or 2-hour PG ≥ 7.8-11.0 mmol/l during 75 gram OGTT
   2. HbA1c ≥ 5.7-6.4%
   3. At least one of the following risk factors:-

      * History of gestational diabetes
      * Family history of diabetes in first degree relative
      * 2 components or more of the metabolic syndrome (triglyceride ≥ 1.7 mmol/L, blood pressure (BP) ≥ 130/80 mmHg, high density-lipoprotein (HDL) cholesterol <1.3 mmol/L in women or <1.1 in men and waist circumference ≥ 80 cm in women or ≥ 90 cm in men). Patients on anti-hypertensive agent for treatment of hypertension or lipid lowering drug for the treatment of hyperlipidaemia will respectively be considered to have one component of the metabolic syndrome.
4. Subject is capable of giving informed consent prior to the initiation of any study related procedures
5. A female subject of childbearing potential who is sexually active with a non-sterilized male partner agrees to use routinely adequate and effective contraception to avoid pregnancy during the study period and up to 30 days after the final visit.
6. The subject is able and willing to consistently record food diary to facilitate CGMS evaluation.

Exclusion Criteria:

1. Subject has received anti-diabetic agents within 6 weeks prior to screening visit.
2. On dietary supplement known to affect glucose or galactose metabolism.
3. History of acute cardiovascular disease including myocardial infarction, acute coronary syndrome or stroke which required hospitalization in the last 12 months.
4. Significant renal impairment with estimated glomerular filtration rate (eGFR) < 60ml/min/1.73m2
5. Known lactose or galactose intolerance.
6. History of eating disorder.
7. Pregnant or lactating female subjects.
8. Subjects with gastrointestinal disease that may interfere with absorption of the investigational product.
9. Subject has received any investigational product within 30 days of randomization visit.
10. Reduced life expectancy or any condition considered by the investigator as unsuitable for enrolment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea OY Luk, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Derived] Luk AOY, Zee BCY, Chong M, Ozaki R, Rausch CW, Chan MHM, Ma RCW, Kong APS, Chow FCC, Chan JCN. A proof-of-concept study to evaluate the efficacy and safety of BTI320 on post-prandial hyperglycaemia in Chinese subjects with pre-diabetes. BMC Endocr Disord. 2018 Aug 31;18(1):59. doi: 10.1186/s12902-018-0288-5. PMID 30170579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the Diabetes and Endocrine Research Centre, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong SAR.
Pre-assignment Details: 77 subjects were screened and 60 subjects met the eligibility criteria to be randomized.
Period: Overall Study
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Started | 24 | 24 | 12
Completed | 22 | 23 | 12
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo | Total
Number analyzed (Participants) | 24 | 24 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (8.6) | 58.5 (8.5) | 57.1 (10.9) | 56.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 9 | 32
  Male | 13 | 12 | 3 | 28
Region of Enrollment [Number; unit: participants]
  Hong Kong | 24 | 24 | 12 | 60
Body weight [Mean (Standard Deviation); unit: kg] | 74.2 (16.9) | 71.0 (16.2) | 63.9 (20.0) | 70.9 (17.4)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 28.0 (5.8) | 26.9 (4.4) | 25.1 (4.3) | 27.0 (5.0)
Waist circumference [Mean (Standard Deviation); unit: cm] | 95.0 (15.6) | 90.6 (9.1) | 88.0 (15.7) | 91.8 (13.5)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121.7 (13.2) | 125.4 (16.2) | 127.8 (8.7) | 124.0 (13.8)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 78.4 (6.8) | 78.7 (7.2) | 80.4 (7.3) | 78.9 (7.0)
Fructosamine [Mean (Standard Deviation); unit: umol/L] | 268.5 (18.3) | 272.2 (20.2) | 278.9 (22.0) | 272.1 (19.9)
HbA1c [Mean (Standard Deviation); unit: %] — Glycated hemoglobin
  % | 6.0 (0.3) | 6.0 (0.3) | 6.1 (0.3) | 6.0 (0.3)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.9 (1.1) | 4.9 (1.0) | 5.3 (0.8) | 5.0 (1.0)
Impaired fasting glucose [Number; unit: participants] | 3 | 1 | 0 | 4
Impaired glucose tolerance [Number; unit: participants] | 10 | 8 | 5 | 23
Impaired fasting glucose and impaired glucose tolerance [Number; unit: participants] | 4 | 7 | 4 | 15
Normal glucose tolerance [Number; unit: participants] | 7 | 8 | 3 | 18
1-hour post-prandial glucose AUC [Mean (Standard Deviation); unit: mmol/L*hour] — 1-hour post-prandial glucose incremental area under curve on continuous glucose monitoring system
  mmol/L*hour | 5.91 (0.53) | 6.22 (0.72) | 6.33 (0.64) | 6.12 (0.65)
2-hour post-prandial glucose AUC [Mean (Standard Deviation); unit: mmol/L*hour] — 2-hour post-prandial glucose incremental area under curve on continuous glucose monitoring system
  mmol/L*hour | 12.68 (1.21) | 13.64 (1.87) | 13.49 (1.43) | 13.22 (1.59)
3-hour post-prandial glucose AUC [Mean (Standard Deviation); unit: mmol/L*hour] — 3-hour post-prandial glucose incremental area under curve on continuous glucose monitoring system
  mmol/L*hour | 18.90 (1.69) | 20.20 (2.59) | 20.20 (2.20) | 19.68 (2.25)
72 hour AUC-180 [Mean (Standard Deviation); unit: mmol/L*hour] — Area under curve for glucose levels >180 mg/dL on continuous glucose monitoring system
  mmol/L*hour | 0.40 (1.85) | 1.71 (3.35) | 2.73 (7.64) | 1.39 (4.17)
Mean blood glucose [Mean (Standard Deviation); unit: mmol/L] — Mean blood glucose on continuous glucose monitoring system
  mmol/L | 6.01 (0.45) | 6.20 (0.63) | 6.45 (0.54) | 6.18 (0.56)
Mean post-meal maximum glucose [Mean (Standard Deviation); unit: mmol/L] — Mean post-meal maximum glucose on continuous glucose monitoring system
  mmol/L | 7.45 (0.75) | 8.20 (1.31) | 8.07 (1.00) | 7.88 (1.09)
Mean amplitude of glucose excursion [Mean (Standard Deviation); unit: mmol/L] — Mean amplitude of glucose excursion on continuous glucose monitoring system
  mmol/L | 2.06 (0.69) | 2.68 (1.01) | 3.21 (3.16) | 2.55 (1.63)
Percentage coefficient of variation [Mean (Standard Deviation); unit: %] — Percentage coefficient of variation on continuous glucose monitoring system
  % | 15.49 (4.43) | 19.07 (6.61) | 18.00 (7.60) | 17.46 (6.20)
Standard deviation [Mean (Standard Deviation); unit: mmol/L] — Standard deviation on continuous glucose monitoring system
  mmol/L | 0.93 (0.28) | 1.19 (0.44) | 1.18 (0.59) | 1.09 (0.43)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Fructosamine in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo
Time Frame: From baseline to Week 4
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 23 | 24 | 12
umol/L | -5.2 (14.1) | -9.4 (8.9) | -8.8 (12.5)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.57, ANCOVA — The p-value of treatment effects relative to placebo was obtained by ANCOVA analysis comparing the outcome values adjusted for age, gender and baseline measurements; Mean Difference (Net) = 2.46, 95% CI 2-sided [-6.28 to 11.20]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.72, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.57, 95% CI 2-sided [-10.3 to 7.11]

2. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean Post-prandial Glucose Incremental Area Under Curve on Continuous Glucose Monitoring System
Description: Changes in 3-hour post-prandial glucose incremental area under curve on continuous glucose monitoring system from baseline to Week 16.
  Note that this is not a pharmacokinetic study and this is not pharmacokinetic data as we are not measuring drug levels. Here we are examining glucose levels after meals as one of the anticipated glycemic outcomes of using glucose-lowering therapy (BTI320 in this case). With data-analysis based on continuous glucose monitoring, it is conventional to present post-prandial (i.e. post-meal) glucose incremental area under curve at up to 3 hours. It is not meaningful to look at post-meal glucose changes at more than 3 hours after meal for the obvious reason that subject might have taken another meal by then.
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L*hour
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L*hour | 0.07 (1.99) | -0.65 (1.93) | -0.68 (1.43)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.66, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.91 to 1.42]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.90, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.07, 95% CI 2-sided [-1.03 to 1.18]

3. Secondary Outcome: Changes in Subjects Treated With Low Dose BTI320 and High Dose BTI320 Compared With Placebo in Mean Post-meal Maximum Glucose on Continuous Glucose Monitoring System
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.13 (0.99) | -0.36 (0.87) | -0.14 (0.58)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.86, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.50 to 0.59]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.59, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.66 to 0.38]

4. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean Amplitude of Glucose Excursion on Continuous Glucose Monitoring System
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 20 | 23 | 12
mmol/L | -0.04 (0.77) | -0.48 (0.88) | -0.92 (3.23)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.62, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.44 to 0.73]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.97, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.52 to 0.55]

5. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean Blood Glucose on Continuous Glucose Monitoring System
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 16 | 22 | 11
mmol/L | -0.01 (0.52) | -0.06 (0.50) | -0.32 (0.56)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.40, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.20 to 0.51]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.49, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.21 to 0.44]

6. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Area Under Curve for Glucose Levels >180mg/dL on Continuous Glucose Monitoring System
Description: Area under curve for glucose levels >180 mg/dL over 72 hours
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L*hour
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 16 | 22 | 11
mmol/L*hour | -0.19 (2.58) | -1.67 (3.51) | -1.38 (9.41)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.41, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.84, 95% CI 2-sided [-2.88 to 1.21]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.15, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.34, 95% CI 2-sided [-3.18 to 0.51]

7. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Standard Deviation of Glucose on Continuous Glucose Monitoring System
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 16 | 22 | 11
mmol/L | -0.09 (0.32) | -0.23 (0.31) | -0.14 (0.68)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.64, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.29 to 0.18]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.41, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.30 to 0.12]

8. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Percent Coefficient of Variation on Continuous Glucose Monitoring System
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: % of coefficient of variation
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 16 | 22 | 11
% of coefficient of variation | -1.6 (4.4) | -3.5 (4.5) | -1.1 (8.8)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.46, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.19, 95% CI 2-sided [-4.43 to 2.05]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.24, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.75, 95% CI 2-sided [-4.72 to 1.21]

9. Secondary Outcome: Changes in HbA1c in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: percent glycated hemoglobin
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
percent glycated hemoglobin | -0.01 (0.19) | -0.02 (0.16) | -0.04 (0.20)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.83, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.13 to 0.10]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.48, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.16 to 0.08]

10. Secondary Outcome: Changes in Fructosamine in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
umol/L | -5.0 (18.6) | -6.8 (12.0) | -9.8 (10.2)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.83, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.14, 95% CI 2-sided [-9.17 to 11.45]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.86, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.92, 95% CI 2-sided [-11.1 to 9.27]

11. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Area Under Curve of Glucose During Standard Meal Tolerance Test From 0 Minute to 120 Minutes
Description: Changes in area under curve of glucose from 0 minute to 120 minutes from baseline to Week 16
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L*minute
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L*minute | -63.6 (103.9) | -24.5 (132.2) | -84.9 (150.4)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.75, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -13.6, 95% CI 2-sided [-99.6 to 72.3]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.34, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 40.0, 95% CI 2-sided [-43.9 to 123.9]

12. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Area Under Curve of Insulin During Standard Meal Tolerance Test From 0 Minute to 120 Minutes
Description: Changes in area under curve of insulin from 0 minute to 120 minutes from baseline to Week 16
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mIU/L*minute
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 22 | 12
mIU/L*minute | -1533.7 (3171.6) | -382.8 (2781.6) | -1225.8 (3922.9)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.23, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -980.0, 95% CI 2-sided [-2604 to 643.8]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.68, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 323.9, 95% CI 2-sided [-1269 to 1916.6]

13. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Area Under Curve of C-peptide During Standard Meal Tolerance Test From 0 Minute to 120 Minutes
Description: Changes in area under curve of C-peptide from 0 minute to 120 minutes from baseline to Week 16
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: ug/L*minute
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 22 | 12
ug/L*minute | -56.2 (193.1) | -22.9 (170.9) | -120.8 (257.8)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.79, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 15.0, 95% CI 2-sided [-99.6 to 129.6]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.29, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 60.1, 95% CI 2-sided [-52.5 to 172.6]

14. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Glucagon-like Peptide 1 During Standard Meal Tolerance Test From 0 Minute to 120 Minutes
Description: Changes in area under curve of glucagon-like peptide-1 from 0 minute to 120 minutes from baseline to Week 16
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: pmol/L*minute
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
pmol/L*minute | 117.0 (340.6) | 130.9 (514.1) | 107.9 (197.4)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.37, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -120.2, 95% CI 2-sided [-385.3 to 144.9]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.69, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 49.0, 95% CI 2-sided [-198.1 to 296.2]

15. Secondary Outcome: Proportion of Subjects With Impaired Fasting Glucose or Impaired Glucose Tolerance in Low Dose BTI320, High Dose BTI320 and Placebo Group
Description: Proportion of subjects with impaired fasting glucose, impaired glucose tolerance, both impaired fasting glucose and impaired glucose tolerance, HbA1c 5.7-6.4%, or type 2 diabetes at 30 days post-treatment
Time Frame: From baseline to 30 days post-treatment
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Number; unit: percentage of subjects
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
percentage of subjects | 100 | 95.7 | 100

16. Secondary Outcome: Changes in Blood Pressures in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Description: Changes in systolic blood pressures from baseline to Week 16
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
mmHg | -0.5 (10.6) | -0.7 (13.5) | -3.5 (15.4)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.57, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.2, 95% CI 2-sided [-9.8 to 5.5]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.79, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.0, 95% CI 2-sided [-6.6 to 8.6]

17. Secondary Outcome: Changes in Waist Circumference in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
cm | -2.5 (3.4) | -1.5 (3.4) | -1.8 (3.6)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.54, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.8, 95% CI 2-sided [-3.4 to 1.8]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.68, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.5, 95% CI 2-sided [-2.0 to 3.1]

18. Secondary Outcome: Changes in Body Weight in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
kg | -1.7 (2.4) | -0.5 (1.9) | -0.1 (1.9)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.03, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.7, 95% CI 2-sided [-3.2 to -0.1]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.86, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.7 to 1.4]

19. Secondary Outcome: Changes in Lipids in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Description: Changes in total cholesterol from baseline to Week 16.
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
mmol/L | -0.0 (0.75) | -0.2 (0.56) | -0.15 (0.65)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.90, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.39 to 0.44]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.30, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.63 to 0.20]

20. Secondary Outcome: Changes in High-sensitivity C-reactive Protein in Subjects Treated With High Dose and Low Dose BTI320 Compared Placebo
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
mg/L | -0.85 (5.78) | 0.09 (2.00) | -0.89 (1.57)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.52, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.62, 95% CI 2-sided [-1.32 to 2.57]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.24, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.13, 95% CI 2-sided [-0.75 to 3.05]

21. Secondary Outcome: Changes in Urate in Subjects Treated With High Dose and Lose Dose BTI320 Compared to Placebo
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
mmol/L | -0.008 (0.054) | 0.006 (0.053) | -0.015 (0.036)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.93, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.002, 95% CI 2-sided [-0.035 to 0.038]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.40, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.015, 95% CI 2-sided [-0.021 to 0.051]

22. Secondary Outcome: Changes in Quality of Life Measures in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Description: Changes in WHOQOL-BREF physical health domain score from baseline to Week 16. This is a sub-scale of the WHOQOL-BREF. Possible scores range from minimal of 4 to maximum of 20. Higher score indicate better physical health domain.
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
units on a scale | -0.6 (1.4) | 0.0 (1.3) | 0.1 (1.1)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.36, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.2 to 0.5]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.36, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.4 to 1.2]

23. Secondary Outcome: Changes in Measures of Food Satiety in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Description: Changes to question of "how full do you feel" in the Appetite Questionnaire adopted from Hill and Blundell from baseline and Week 16. Scale score ranges from minimum of 0 to maximum of 10. 10 being the most full and 0 being the least full.
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
units on a scale | -0.4 (2.7) | 1.0 (3.2) | 1.3 (2.6)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.09, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.82, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group

24. Secondary Outcome: Changes in Measures of Nutritional Intake in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Description: Changes in daily calories intake from baseline to Week 16
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
kcal | -237.4 (358.8) | -75.0 (486.2) | -320.9 (794.8)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.68, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.26, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group

25. Secondary Outcome: Changes in Measures of Exercise in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Description: Changes in the number of days per week that the subject spent walking for at least 10 minutes from baseline to Week 16
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 22 | 12
Days | -0.1 (1.7) | -0.5 (2.1) | 0.2 (0.6)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.67, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.30, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group

26. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean 1 Hour Post-prandial Glucose Incremental Area Under Curve on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L*hour
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L*hour | 0.11 [-0.18 to 0.41] | -0.07 [-0.33 to 0.19] | -0.15 [-0.49 to 0.20]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — The p-value of treatment effects (reference to placebo) were obtained by mixed effect model analysis comparing the outcome values adjusted with repeated measures, ages and gender; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.48 to -0.11]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.32 to 0.04]

27. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean 2 Hour Post-prandial Glucose Incremental Area Under Curve on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L*hour
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L*hour | 0.08 [-0.62 to 0.78] | -0.51 [-1.10 to 0.08] | -0.31 [-0.92 to 0.31]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.59, 95% CI 2-sided [-1.01 to -0.18]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.42, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.57 to 0.24]

28. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean 3 Hour Post-prandial Glucose Incremental Area Under Curve on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L*hour
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L*hour | 0.14 [-0.85 to 1.14] | -0.68 [-1.51 to 0.14] | -0.69 [-1.59 to 0.21]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.74, 95% CI 2-sided [-1.35 to -0.14]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.57, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.75 to 0.42]

29. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in 1 Hour Post-prandial Mean Blood Glucose on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.12 [-0.20 to 0.44] | -0.08 [-0.36 to 0.20] | -0.16 [-0.53 to 0.22]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.52 to -0.12]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.14, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.34 to 0.05]

30. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in 2 Hour Post-prandial Mean Blood Glucose on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.12 [-0.24 to 0.48] | -0.19 [-0.49 to 0.11] | -0.08 [-0.42 to 0.26]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.31, 95% CI 2-sided [-0.52 to -0.10]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.38, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.30 to 0.12]

31. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in 3 Hour Post-prandial Mean Blood Glucose on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.15 [-0.19 to 0.48] | -0.14 [-0.40 to 0.12] | -0.04 [-0.34 to 0.25]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.48 to -0.07]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.41, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.28 to 0.11]

32. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean Blood Glucose During 24 Hours on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | -0.05 [-0.27 to 0.17] | -0.05 [-0.26 to 0.16] | -0.16 [-0.38 to 0.06]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.40 to 0.03]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.38 to 0.03]

33. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Post-prandial Maximum Glucose on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.15 [-0.34 to 0.64] | -0.38 [-0.75 to 0.00] | -0.14 [-0.51 to 0.23]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.39, 95% CI 2-sided [-0.67 to -0.12]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.54, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.35 to 0.18]

34. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Mean Post-prandial Maximum Glucose During 24 Hours on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.10 [-0.38 to 0.58] | -0.52 [-0.91 to -0.12] | -0.35 [-0.82 to 0.12]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.81 to -0.03]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.63, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.48 to 0.29]

35. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Standard Deviation of Blood Glucose During 1 Hour Post-prandial on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.00 [-0.15 to 0.15] | -0.18 [-0.31 to -0.05] | -0.05 [-0.19 to 0.09]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.13 to 0.02]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.73, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.06 to 0.09]

36. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Standard Deviation of Blood Glucose During 2 Hours Post-prandial on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.02 [-0.12 to 0.16] | -0.13 [-0.25 to 0.00] | -0.01 [-0.13 to 0.11]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.15 to 0.00]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.46, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.05 to 0.10]

37. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Standard Deviation of Blood Glucose During 3 Hours Post-prandial on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | 0.01 [-0.13 to 0.15] | -0.12 [-0.23 to -0.01] | -0.02 [-0.14 to 0.09]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.15 to 0.00]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.46, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.05 to 0.10]

38. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Standard Deviation of Blood Glucose Over 24 Hours on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
mmol/L | -0.05 [-0.20 to 0.10] | -0.20 [-0.33 to -0.07] | -0.18 [-0.61 to 0.25]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.31 to -0.02]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.87, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.13 to 0.15]

39. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Percent Coefficient of Variation of Blood Glucose Over 1 Hour Post-prandial on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: % of coefficient of variation
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
% of coefficient of variation | -0.26 [-1.99 to 1.47] | -2.46 [-4.03 to -0.90] | -0.60 [-2.18 to 0.98]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.34, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.48, 95% CI 2-sided [-1.46 to 0.50]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.64, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.73 to 1.18]

40. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Percent Coefficient of Variation of Blood Glucose Over 2 Hours Post-prandial on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: % of coefficient of variation
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
% of coefficient of variation | -0.06 [-1.54 to 1.42] | -1.28 [-2.71 to 0.16] | -0.01 [-1.67 to 1.65]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.62, 95% CI 2-sided [-1.50 to 0.26]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.46 to 1.24]

41. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Percent Coefficient of Variation of Blood Glucose Over 3 Hours Post-prandial on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: % of coefficient of variation
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
% of coefficient of variation | -0.18 [-1.73 to 1.38] | -1.37 [-2.67 to -0.08] | -0.33 [-1.93 to 1.27]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.62 to 0.31]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.42, 95% CI 2-sided [-0.51 to 1.36]

42. Secondary Outcome: Changes in Subjects Treated With Low Dose and High Dose BTI320 Compared With Placebo in Percent Coefficient of Variation of Blood Glucose Over 24 Hours on Continuous Glucose Monitoring System Repeated Measures Analysis
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (95% Confidence Interval); unit: % of coefficient of variation
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 21 | 23 | 12
% of coefficient of variation | -0.84 [-2.99 to 1.31] | -3.04 [-4.95 to -1.13] | -2.68 [-10.09 to 4.73]
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -2.14, 95% CI 2-sided [-4.36 to 0.09]
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.69, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 0.43, 95% CI 2-sided [-1.71 to 2.58]

43. Other Pre Specified Outcome: Changes in Serum Creatinine in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Time Frame: From baseline to Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
umol/L | -4.3 (7.0) | -3.5 (8.5) | -7.0 (6.7)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.29, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.22, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group

44. Other Pre Specified Outcome: Changes in Measures of Liver Function in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Time Frame: From baseline to Week 4, Week 8, Week 12, and Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
IU/L | 2.6 (12.5) | 1.4 (8.5) | -0.9 (10.2)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.41, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.48, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group

45. Other Pre Specified Outcome: Changes in Complete Blood Count in Subjects Treated With High Dose and Low Dose BTI320 Compared to Placebo
Time Frame: From baseline to Week 4, Week 8, Week 12, and Week 16
Population: Intention to treat, as defined by all subjects who have received at least one dose of BTI320
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Number analyzed (Participants) | 22 | 23 | 12
g/dL | -0.3 (0.4) | -0.4 (0.5) | -0.4 (0.4)
Statistical Analysis 1: Comparison: BTI320 4 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.61, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group
Statistical Analysis 2: Comparison: BTI320 8 Grams vs BTI320 Matching Placebo; Test type: Superiority or Other; p = 0.89, t-test, 2 sided — The univariate p-value of treatment group was obtained by t-tests comparing the changes to that of placebo group

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | BTI320 4 Grams | BTI320 8 Grams | BTI320 Matching Placebo
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 18/24 | 16/24 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTI320 4 Grams (N=24) | BTI320 8 Grams (N=24) | BTI320 Matching Placebo (N=12)
High grade osteosarcoma at left distal femur (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTI320 4 Grams (N=24) | BTI320 8 Grams (N=24) | BTI320 Matching Placebo (N=12)
Abdominal distension (Gastrointestinal disorders) | 6 (8) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (6) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 7 (7) | 8 (8) | 2 (2)
Frequent bowel movements (Gastrointestinal disorders) | 4 (4) | 2 (2) | 5 (5)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tooth fracture (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No